CLINICAL TRIAL: NCT03405480
Title: Pulmonary Rehabilitation to Improve Physical Capacity After Pulmonary Embolism - a Randomized Controlled Trial - The REHAB Study
Brief Title: Pulmonary Rehabilitation to Improve Physical Capacity After Pulmonary Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: University Hospital, Akershus (Other); Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/1940 (REK)
Record Dates: First submitted 2018-01-11; First posted 2018-01-23 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Dyspnea; Post Pulmonary Embolism Syndrome; PPS; Rehabilitation; Cardiac magnetic resonance imaging (CMR)
MeSH Terms: conditions — Pulmonary Embolism; Dyspnea | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation (Experimental): Physiotherapist-supervised outpatient rehabilitation program 2 times a week for a total of 8 weeks.
  Interventions: Other: Rehabilitation
- No rehabilitation (No Intervention): Patients will receive usual care, including information pamphlets with information on the disease and the general importance of exercise.

INTERVENTIONS:
Other: Rehabilitation — Rehabilitation
  Arms: Rehabilitation

SUMMARY:
This project aims to evaluate a rehabilitation program as treatment and uncover potential pathophysiological mechanisms of a newly identified chronic condition named "Post Pulmonary Embolism Syndrome" (PPS).

DETAILED DESCRIPTION:
The newly identified Post Pulmonary Embolism Syndrome (PPS) is characterized by chronic persistent, but unexplained dyspnea (i.e. without signs of pulmonary hypertension or pulmonary abnormality). Symptoms are considerable, but less severe than in CTEPH patients. A recent study performed by our group confirmed that up to 50% of our patients complained of various grades of persistent unexplained dyspnea 1-10 years after the diagnosis of PE.

In this multifaceted project we wish to evaluate the effect of an eight week rehabilitation program led and supervised by a trained physiotherapist on exercise capacity in PPS patients. This interventional part of the study will be formed as a randomized controlled trial. Patients will be randomized to either usual care or a physiotherapist-supervised rehabilitation program.

The study also aims to explore potential underlying pathophysiological mechanisms in PPS, using state of the art methods such as cardiac magnetic resonance imaging and transthoracic echocardiography involving novel methods focusing on the right ventricle. The pathophysiological part of the study will be formed as a case control study, where post PE-patients who do not fulfill the criteria for PPS will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Objectively diagnosed symptomatic pulmonary embolism by CTPA or high-probability scintigraphy 6 months to 6 years before inclusion
* Persistent dyspnea defined as modified Medical Research Council (mMRC) breathlessness scale >= 1 that has appeared or worsened after the diagnosis of PE (eligibility criteria for randomization)

Exclusion Criteria:

* Significant pulmonary disease (COPD GOLD >= 2, restrictive pulmonary disease, lung cancer or pleural disease.
* Heart failure (either HFrEF, HFmrEF or HFpEF as defined in ESC guidelines)
* Significant valvular heart disease
* Chronic thromboemboli pulmonary hypertension (CTEPH)
* Patients unfit for rehabilitation or walking tests du to old age, physical disability or disease
* Patients with a history of poor compliance or any condition that would interfere with the ability to comply with the study protocol e.g. history of drug abuse, excessive alcohol beverage consumption, cognitive dysfunction or severe psychiatric disease
* Active malignancy
* Life expectancy less than 3 months
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
ISWT | ISWT wil be performed at 12 weeks and 36 weeks after baseline
  Change in "Incremental Shuttle Walk Test" will be primary endpoint for interventional part of the study

SECONDARY OUTCOMES:
mMRC | 12 weeks and 36 weeks after inclusion
  The effect of rehabilitation on dyspnea measured by mMRC breathlessness scale
Sensewear | 12 weeks and 36 weeks after baseline
  The effect of PRP on daily physical activity as measured with an activity monitor (Sensewear)
HRQoL by EQ-5d | 12 weeks and 36 weeks after baseline
  The effect of rehabilitation on HRQoL measured by EQ-5D
HRQoL by PEmb-QoL | 12 weeks and 36 weeks after baseline
  The effect of rehabilitation on HRQoL measured by PEmb-QoL
Long term effect of physical capacity | 6 months after completing rehabilitation
  The long-term effect of rehabilitation on physical capacity measured by ISWT, 6 months after completing the rehabilitation
Test-retest reliability of the ISWT in this patient population | At baseline, 12 weeks and 36 weeks
  Test-retest reliability of the ISWT in this patient population
Minimum clinically important difference for ISWT | 36 weeks after baseline
  Establish the minimum clinically important difference (MID) for the ISWT in patients with PPS expressed in meters.
Proportion of patients who achieves the established minimum clinically important difference | 36 weeks after baseline
  Proportion of patients who achieves the established minimum clinically important difference for ISWT for this population

OTHER OUTCOMES:
Myocardial fibrosis evaluated by cardiac MRI | At baseline
  The primary objective in the pathophysiology part of the study is to investigate whether diffuse myocardial fibrosis shown by CMR is associated with PPS

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, MD. Assoc.Prof, Study Director — Hospital of Østfold, Kalnes
Locations (1):
- The hospital of Østfold, Kalnes, Grålum, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhayyat A, Stavem K, Jervan O, Hilde JM, Rashid D, Gleditsch J, Ghanima W, Steine K. Stress Echocardiography to Detect Exercise Pulmonary Hypertension in Patients With Chronic Thromboembolic Pulmonary Disease. Pulm Med. 2026 Jan 28;2026:4127338. doi: 10.1155/pm/4127338. eCollection 2026. PMID 41623859
- [Derived] Jervan O, Haukeland-Parker S, Gleditsch J, Tavoly M, Klok FA, Steine K, Johannessen HH, Spruit MA, Atar D, Holst R, Astrup Dahm AE, Sirnes PA, Stavem K, Ghanima W. The Effects of Exercise Training in Patients With Persistent Dyspnea Following Pulmonary Embolism: A Randomized Controlled Trial. Chest. 2023 Oct;164(4):981-991. doi: 10.1016/j.chest.2023.04.042. Epub 2023 May 5. PMID 37149257
- [Derived] Fabyan KD, Holley AB. Postpulmonary embolism syndrome. Curr Opin Pulm Med. 2021 Sep 1;27(5):335-341. doi: 10.1097/MCP.0000000000000789. PMID 34127618
- [Derived] Haukeland-Parker S, Jervan O, Johannessen HH, Gleditsch J, Stavem K, Steine K, Spruit MA, Holst R, Tavoly M, Klok FA, Ghanima W. Pulmonary rehabilitation to improve physical capacity, dyspnea, and quality of life following pulmonary embolism (the PeRehab study): study protocol for a two-center randomized controlled trial. Trials. 2021 Jan 6;22(1):22. doi: 10.1186/s13063-020-04940-9. PMID 33407792